CLINICAL TRIAL: NCT03317483
Title: The Comprehensive Analysis of Efficacy and Safety of CalliSpheres® Drug-eluting Beads Transarterial Chemoembolization in 367 Patients With Liver Cancer: a Multiple-center Cohort Study (CTILC Study)
Brief Title: DEB-TACE Treatment in 367 Liver Cancer Patients
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, guoliang shao, Vice president of Zhejiang Cancer Hospital, Zhejiang Cancer Hospital
Other Study IDs: CTILC
Record Dates: First submitted 2017-10-13; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 404 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction:The drug-eluting beads transarterial chemoembolization (DEB-TACE) is introduced to better improve efficacy and reduce the systemic toxicity in liver cancer patients on account of its higher intratumoral chemotherapeutic drug concentration and reduced drug infiltration into systemic circulation. This study aimed to investigate the efficacy, safety and prognostic factors of DEB-TACE treatment in Chinese patients with liver cancer.

Hypothesis:DEB-TACE illustrates a better treatment response, progression free survival (PFS), overall survival (OS) and less common adverse events (AEs) in liver cancer patients.

Objective: to investigate the efficacy, safety and prognostic factors of DEB-TACE treatment in Chinese patients with liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as primary HCC, primary ICC or secondary liver cancer confirmed by pathological findings, clinical features or radiographic examinations according to American Association for the Study of the Liver Diseases (AASLD) guidelines;
2. Age above 18 years;
3. About to receive DEB-TACE treatment with CalliSpheres® according to clinical needs and patients' willing.
4. Able to be followed up regularly;
5. Life expectancy above 12 months.

Exclusion Criteria:

1. History of liver transplantation;
2. History of hematological malignances;
3. Severe hepatic failure or renal failure;
4. Contraindication for angiography, embolization procedure or artery puncture;
5. Patients with cognitive impairment, or unable to understand the study consents.
6. Women in gestation or lactation period.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 367 liver cancer patients about to receive DEB-TACE treatment from 2015/11/12 to 2016/11/04 were prospectively included in CTILC study.
Sampling Method: Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Treatment response | One-three months after DEB-TACE treatment
  Treatment response was assessed at 1-3 months after DEB-TACE treatment according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) by enhanced computerized tomography (CT) or magnetic resonance imaging (MRI) examination.

SECONDARY OUTCOMES:
overall survival | The median follow-up duration was 171 (range from 38 to 404) days.
  OS was calculated from the time of DEB-TACE operation to the time of patient's death from any causes.
Liver function evaluation | One week post and 1-3 months post DEB-TACE treatment.
  Liver function indexes including ALB, TP, TBIL, TBA, ALT, AST and ALP were recorded before, 1 week post and 1-3 months post DEB-TACE treatment to evaluate the influence of DEB-TACE on liver function. The analysis of liver function evaluation was based on the treatment records of DEB-TACE .
Adverse events (AEs) | During DEB-TACE operation and 1 month after DEB-TACE operation.
  AEs were recorded during DEB-TACE operation and 1 month after DEB-TACE operation, and the analysis of AEs was based on the treatment records of DEB-TACE.

REFERENCES:
- [Derived] Luo J, Zheng J, Shi C, Fang J, Peng Z, Huang J, Sun J, Zhou G, Li T, Zhu D, Xu H, Hou Q, Ying S, Sun Z, Du H, Xie X, Cao G, Ji W, Han J, Gu W, Guo X, Shao G, Yu Z, Zhou J, Yu W, Zhang X, Li L, Hu H, Hu T, Wu X, Chen Y, Ji J, Hu W. Drug-eluting beads transarterial chemoembolization by CalliSpheres is effective and well tolerated in treating intrahepatic cholangiocarcinoma patients: A preliminary result from CTILC study. Medicine (Baltimore). 2020 Mar;99(12):e19276. doi: 10.1097/MD.0000000000019276. PMID 32195932